CLINICAL TRIAL: NCT03420352
Title: Serum Blood Clotting Changes During Blood Sampling Via Non-luer One-way Filter Valve Intravenous Needle: Implication on the Epidural Blood Patch Procedure
Brief Title: Non-Luer Butterfly Needle With One-way Valve for the Epidural Blood Patch: Does it Alter Blood Clotting?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 196031
Record Dates: First submitted 2018-01-19; First posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Post-Dural Puncture Headache; Low Pressure Headache
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Thrombelastography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- butterfly needle with valve (Other): thromboelastography
  Interventions: Diagnostic Test: Thromboelastography
- Standard hypodermic needle (Other): thromboelastography
  Interventions: Diagnostic Test: Thromboelastography

INTERVENTIONS:
Diagnostic Test: Thromboelastography — paired TEG analysis undertaken from participants with the two different needles

SUMMARY:
The Department of Health recommends using equipment which prevents wrong route drug administration. However, the epidural blood patch requires equipment that connects to the intravenous and epidural route. To comply with these recommendations a non-Luer butterfly needle with one-way valve has been produced. The one-way valve and length of tubing has the potential to activate the clotting cascade. This could reduce the time clinicians have to utilise the blood in the syringe. Also any alteration in clotting could affect the therapeutic value of the epidural blood patch. The primary objective of this research was to determine if phlebotomy using this new 21G needle altered blood clotting, determined by thromboelastograph analysis, compared to a standard 21G hypodermic needle.

DETAILED DESCRIPTION:
Ethical approval was gained from the Health Research Authority (North West - Greater Manchester South Research Ethics Committee, REC Reference Number: 16/NW/0570). After informed consent, we enrolled participants

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female.
* Aged 18 years or above.
* Within first 2 days postnatal for postnatal group
* Healthy participants must be in good health.
* Able (in the Investigators opinion) and willing to comply with all study requirements.
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the study.

Exclusion Criteria:

* Any medical condition
* In postnatal group, women with haemorrhage greater than 1L
* In postnatal group, less than 12 hours post prophylactic dalteparin
* Any clotting abnormality
* On any medication including herbal medication (vitamins taken during pregnancy are acceptable)
* Age less than 18 years at recruitment
* Adults who are not capable of giving valid consent
* Adults with learning disabilities/ difficulties
* Adults in emergency situations
* Unable to speak or read English
* Prisoners
* Adults unable to consent for themselves
* Any person considered to have a particularly dependent relationship with investigators
* Any others deemed to belong to a vulnerable group.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* Participants who have participated in another research study involving an investigational product in the past 12 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-04-28 (Actual); Study Completion 2017-04-28 (Actual)

PRIMARY OUTCOMES:
Reaction Time (R-time) (Minutes) | 1 hour
  We will measure the thromboelastography (TEG) results of the patients blood with each needle. The TEG analysis will provide us with the R-time
Maximum amplitude (millimetre) (MA) | 1 hour
  We will measure the thromboelastography (TEG) results of the patients blood with each needle. The TEG analysis will provide us with the MA
Lysis-30 (%) (LY30) | 1 hour
  We will measure the thromboelastography (TEG) results of the patients blood with each needle. The TEG analysis will provide us with the LY30

CONTACTS AND LOCATIONS:
Overall Officials: Asif Mahmood, MBChB,FRCA, Principal Investigator — University Hospital Leicester
Locations (1):
- University Hospital Leicester, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified data with all primary outcomes measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From publication of paper, for as long as required
Access Criteria: Data access requests will be reviewed by an external independent review panel. Requesters will be required to sign a data access agreement.

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2017-01-01): https://cdn.clinicaltrials.gov/large-docs/52/NCT03420352/Prot_SAP_000.pdf
  • Informed Consent Form: healthy volunteer consent (2016-11-15): https://cdn.clinicaltrials.gov/large-docs/52/NCT03420352/ICF_001.pdf
  • Informed Consent Form: Pregnant volunteer consent (2016-07-30): https://cdn.clinicaltrials.gov/large-docs/52/NCT03420352/ICF_002.pdf